CLINICAL TRIAL: NCT06867848
Title: Augmentation of Facial Wall in Defective Fresh Extraction Site for Immediate Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuhayra Ashour Muhammed (Other Government)
Responsible Party: Sponsor-Investigator, Nuhayra Ashour Muhammed, candidate of master degree in faculty of dental medicine for girls, Faculty of Dental Medicine for Girls
Organization: Faculty of Dental Medicine for Girls (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OR SUR-102-1-E
Record Dates: First submitted 2025-01-05; First posted 2025-03-10 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-03

CONDITIONS: the Augmentation of Labial Defective Wall in Fresh Extraction Socket
Keywords: labial bone augmentation, immediate implant placement .; laminar bone membrane effect; pericardium membrane effect

STUDY DESIGN:
Intervention Model Description: the study is interventional study containing two groups, each group receiving deferent type of treatment for their result comparison.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- laminar bone membrane (Experimental): hopeless tooth extraction then immediate implant placed , then by using vestibular incision placing laminar bone membrane under the mucogingival tunnel and fill the gap between the laminar bone membrane and the implant with sticky bone
  Interventions: Procedure: laminar bone membrane for labial bone augmentation
- pericardium membrane (Experimental): hopeless tooth extraction then immediate implant placed , then by using vestibular incision placing pericardium membrane under the mucogingival tunnel and fill the gap between the pericardium membrane and the implant with sticky bone
  Interventions: Procedure: laminar bone membrane for labial bone augmentation

INTERVENTIONS:
Procedure: laminar bone membrane for labial bone augmentation — adding laminar bone membrane in one group and pericardium membrane in another group with sticky bone by using vestibular incision in both groups to augment the labial bone over dental implant
  Other Names: pericardium membrane for labial bone augmentation

SUMMARY:
The study is performed to clinically and radiographically assess the efficacy of using enriched bone graft combined with slowly resorbable membrane on bone quality in immediate implant placement in extraction socket in cases with localized facial bone defect.

DETAILED DESCRIPTION:
The study is include twelve participants , and the patients are in rolled in two groups, group one receive implant, sticky bone and laminar bone membrane . group two receive implant, sticky bone and pericardium membrane using vestibular incision and 6 months post operative radiographically assessment is performed to measure labial bone quantity formed .

ELIGIBILITY:
Inclusion Criteria:

* patient with a single hopeless tooth in maxillary anterior region.
* sufficient bone apically and palatally
* presence of natural contralateral tooth for the tooth being replaced
* systemic healthy patients

Exclusion Criteria:

* extraction socket type III
* acute infection in hopeless tooth
* a heavy smoker patient
* pregnant
* had received chemotherapy or radiotherapy in previous year

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
primary stability of implant in Newton centimeter and soft tissue healing | one week postoperative
  Dental implant ratchet to show implant stability and Pink esthetic score for soft tissue healing measurement

SECONDARY OUTCOMES:
labial bone thickness formation in millimeters | 6 months postoperative
  Cone beam computed tomography to show labial bone thickness

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dental medicine for girls, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No